CLINICAL TRIAL: NCT03428009
Title: Dystonia Genotype-Phenotype Correlation: A Study to Identify Additional Genetic Associations That Contribute to Specific Dystonic Phenotypes
Brief Title: Dystonia Genotype-Phenotype Correlation
Status: Recruiting | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jeff Waugh, MD, PhD, Associate Professor, University of Texas Southwestern Medical Center
Other Study IDs: STU 122017-069
Record Dates: First submitted 2018-02-02; First posted 2018-02-09 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Dystonia; Dystonia; Idiopathic; Dystonia, Primary; Dystonia, Secondary; Dystonia, Familial; Dystonia Disorder; Dystonias, Sporadic; Dystonia; Orofacial; Dystonia Lenticularis; Dystonia, Paroxysmal; Dystonia 6; Dystonia 5; Dystonia 8; Dystonia 9; Dystonia 19; Dystonia 10; Dystonia 11; Dystonia 20; Dystonia 12; Dystonia, Focal; Dystonia of Head; Dystonia, Diurnal
Keywords: Dystonia; Control; Magnetic Resonance Imagine; Genotype; Phenotype
MeSH Terms: conditions — Dystonia; Dystonic Disorders; Dystonia 6, torsion; Dystonia, Dopa-responsive; Paroxysmal nonkinesigenic dyskinesia; Choreoathetosis-Spasticity, Episodic; Episodic Kinesigenic Dyskinesia 2; Familial paroxysmal dystonia; Myoclonic dystonia; Paroxysmal Nonkinesigenic Dyskinesia 2; Dystonia 12 | interventions — Magnetic Resonance Spectroscopy; Blood Specimen Collection; Genetic Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Investigators will be collecting blood samples once ( two 8.5 mL Vacutainer tubes) at the participants first study visit to be sent to MGH for genetic analysis. Investigators will aliquot the whole blood collected into cyrovials and ship them overnight on dry ice to the MGH tissue culture bank to be stored and processed. No identifiable information will be sent with the blood samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Dystonia group: Both groups will have blood drawn, undergo clinical assessments, the collection of medical and family history, and an Magnetic Resonance Imaging. This is an observational study and there is no intervention.
  Interventions: Other: Magnetic Resonance Imaging
- Control Group: Both groups will have blood drawn, undergo clinical assessments, the collection of medical and family history, and an Magnetic Resonance Imaging. This is an observational study and there is no intervention.
  Interventions: Other: Magnetic Resonance Imaging

INTERVENTIONS:
Other: Magnetic Resonance Imaging — Study interventions are minimal risk.
  Other Names: Blood Draw for Genetic testing; Clinical Assessments

SUMMARY:
The purpose of this study is to (1) investigate the effect of known dystonia-causing mutations on brain structure and function, to (2) identify structural brain changes that differ between clinical phenotypes of dystonia, and to (3) collect DNA, detailed family history, and clinical phenotypes from patients with idiopathic dystonia with the goal of identifying new dystonia-related genes. Investigators will be recruiting both healthy control subjects and subjects with any form of dystonia. For this study there will be a maximum of two study visit involving a clinical assessment, collection of medical and family history, task training session, an MRI using the learned tasks, and finally a blood draw for genetic analysis. In total, these visits will take 3-5 hours. If the dystonia subjects receive botulinum toxin injections for treatment, the participants and their matched controls will be asked to come for a second visit.

DETAILED DESCRIPTION:
1. Identify a cohort of individuals with known dystonia-related gene mutations, and individuals with idiopathic but presumed-genetic dystonia. Some of these individuals may receive botulinum toxin injections to treat their dystonia per standard of care; in these patients, investigators will image before and after injections to assess for imaging correlates of treatment response.
2. Analyze DNA samples from both the dystonia and healthy individual cohorts to detect the presence of mutations and/or polymorphisms in genes associated with dystonia
3. Collect systematic clinical information, including Tsui Torticollis, Burke-Fahn-Marsden, Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS), Voice Disability Index, Unified Myoclonus Rating Scale, Beck Depression Inventory, Beck Anxiety Inventory and Spielberg Trait Anxiety scales. Scales will be tailored to the type of dystonia, as determined by the clinician referring into the study (i.e., torticollis scales will only be performed on patients with cervical dystonia).
4. Use functional MRI (fMRI), diffusion tensor imaging (DTI), and structural MRI to a) analyze brain activity and structure pre- and post-botulinum toxin injections, b) determine how different stages of movement (execution, preparation, sequencing) influence dystonia and the underlying neural mechanisms, c) identify structural abnormalities shared between clinical sub-types of dystonia. As new MR imaging methods are introduced that may improve the investigators ability to identify or distinguish these abnormalities, the investigator will incorporate these novel sequences into the imaging protocol.
5. Correlate brain activity and structural data with ratings of dystonia severity, location of dystonia, genetic status, and response to treatment (medications and/or botulinum toxin injections).
6. Correlate polymorphism data with dystonia severity, response to botulinum toxin, depression/anxiety severity, and brain activity/structure.

ELIGIBILITY:
General Exclusion (both Dystonia and Control groups):

* Metal in any part of the body (including metal injury to the eye) OR carrying a medical device incompatible with MRI (e.g., metal implants such as surgical clips or pacemakers) OR positive screening per UTSW MRI screening form
* Claustrophobia
* Non-fluent English
* Weight incompatible with MRI safety
* History of head trauma with neurological sequelae, including multiple concussions and/or history of stroke
* Pregnancy
* Serious medical illness or history of serious medical illness, including cancer that was treated with radiation or chemotherapy, heart attack, or a known history of HIV-1 + status
* Subjects with Hepatitis C (by Hepatitis C+ titer)
* Subjects with insulin dependent diabetes mellitus (IDDM)
* Severe respiratory compromise
* In the opinion of the investigator, not able to safely participate in this study

Inclusion Criteria:

* Dystonia group

Previous diagnosis of dystonia which include but is not limited to:

* cervical dystonia (50 subjects)
* blepharospasm (25 subjects)
* limb dystonia (50 subjects)
* spasmodic dysphonia (25 subjects)
* segmental dystonia
* multi-focal dystonia
* Any childhood-onset dystonia (25 subjects) Age > 11 years

  * Control group:

No prior dystonia diagnosis (175 subjects) Age > 11 years

Exclusion Criteria:

* Dystonia group Prior history of or concurrent neurological or psychiatric diagnosis - depression and/or anxiety accepted Current use of non-dystonia neuroactive medications - SSRI/medication for depression and/or anxiety accepted Current use of cervical brace designed for dystonia treatment Prior structural brain injury

Control group:

History of or current neurological or psychiatric diagnosis - depression and/or anxiety accepted, but must not be in active phase Current use of any neuroactive medication, SSRI/medication for depression and/or anxiety accepted

Min Age: 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Investigators will recruit both healthy participants and individuals diagnosed with dystonia of any form for this study. Each Dystonia subject will be matched 1:1 with an unrelated control subject based on: 1) age, +/- 3 years (adults), +/- 1 year (16-18y), +/- 6 months (11-15y); 2) handedness, as determined by the Edinburgh Handedness Inventory, 3) gender, and 4) self-identified racial or ethnic background.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Structural or functional imaging of dystonia and control groups | 3-5 hours at each study visit
  Identify structural or functional imaging measures that distinguish (a) dystonia patients from matched controls, (b) between clinically-defined forms of dystonia
Genetic Analysis of dystonia and control groups | 30 min
  Identify polymorphisms in genes known to cause dystonia that affect the structural or functional imaging measures in dystonia patients and to identify new genes associated with dystonia.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Data and/or sample collection was specifically for research and subjects indicated that their data could be shared with other scientists. Investigators will only send coded data and/or samples with no identifying information. In addition, all whole blood for DNA samples collected for this protocol will be sent for DNA sequencing and genetic analysis at Massachusetts General Hospital in Dr. Nutan Sharma's lab. In addition at Massachusetts General Tissue Culture Core in the Dystonia Partners Research Biobank investigators will contribute the subject's deidentified DNA sample from this protocol for use in future genetic research regarding dystonia.
Time Frame: DNA samples will be stored indefinitely